CLINICAL TRIAL: NCT03274271
Title: A Parallel-group Randomized Trial to Compare the Efficacy of Different Behaviour Change Techniques in the e- and M-health Intervention 'MyPlan 2.0'
Brief Title: Efficacy of Different Behaviour Change Techniques in MyPlan 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: MyPlan2.0
Record Dates: First submitted 2017-06-20; First posted 2017-09-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Disease, Chronic
Keywords: physical activity; sedentary behaviour; eHealth; mHealth; self-regulation; behaviour change techniques; action planning; coping planning; self-monitoring; prevention
MeSH Terms: conditions — Chronic Disease; Motor Activity; Self-Control | interventions — Blood Glucose Self-Monitoring; Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Intervention Model Description: 2x2x2 design with 3 behaviour change techiques provided or not provided
Who Masked: Participant
Masking Description: The different participants will receive different website links to the intervention website, according to their group. The link will not provide information about their group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- AP+CP+M (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with all three behaviour change techniques of interest: action planning (AP), coping planning (CP) and self-monitoring (M).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Action planning; Behavioral: Coping planning; Behavioral: Self-monitoring; Behavioral: Feedback and tips
- AP+CP (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with two of the behaviour change techniques of interest: action planning (AP) and coping planning (CP).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Action planning; Behavioral: Coping planning; Behavioral: Feedback and tips
- AP+M (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with two of the behaviour change techniques of interest: action planning (AP) and self-monitoring (M).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Action planning; Behavioral: Self-monitoring; Behavioral: Feedback and tips
- CP+M (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with two of the behaviour change techniques of interest: coping planning (CP) and self-monitoring (M).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Coping planning; Behavioral: Self-monitoring; Behavioral: Feedback and tips
- M (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with only one of the behaviour change techniques of interest: self-monitoring (M).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Self-monitoring; Behavioral: Feedback and tips
- CP (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with only one of the behaviour change techniques of interest: coping planning (CP).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Coping planning; Behavioral: Feedback and tips
- AP (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' with only one of the behaviour change techniques of interest: action planning (AP).
  They will also receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Action planning; Behavioral: Feedback and tips
- Control (Active Comparator): Participants will receive the e- and mHealth intervention 'MyPlan 2.0' without the three behaviour change techniques of interest (action planning, coping planning, self-monitoring). They will receive general tips and tricks and other behaviour change techniques included in the intervention: tailored feedback and eliciting social support.
  Interventions: Behavioral: Feedback and tips

INTERVENTIONS:
Behavioral: Action planning — Action planning is the behaviour change technique used to make users specify their goal (what they are going to do, when, where, ...).
  Arms: AP; AP+CP; AP+CP+M; AP+M
Behavioral: Coping planning — Coping planning is the behaviour change technique used to make users think about possible hindrances and according solutions when trying to reach their goal.
  Arms: AP+CP; AP+CP+M; CP; CP+M
Behavioral: Self-monitoring — Self-monitoring is the behaviour change technique used to make users keep track of their goal.
  Arms: AP+CP+M; AP+M; CP+M; M
Behavioral: Feedback and tips — In this intervention, users receive tailored feedback on their current health behaviour and tips and tricks to reach their goals. This tips and tricks include the behaviour change technique 'eliciting social support'.

SUMMARY:
The aim of this study is to investigate the effectiveness of intervention 'MyPlan 2.0' and the efficacy of the different behaviour change techniques that are included. Eight groups will be created that will receive a different version of the intervention, varying in three behaviour change techniques (action planning, coping planning, self-monitoring).

DETAILED DESCRIPTION:
The effectiveness of the self-regulation-based e- and m-health intervention 'MyPlan 2.0' on changing physical activity and sedentary behaviour in the adult population will be investigated. Furthermore, the role of three different behaviour change techniques (action planning, coping planning, self-monitoring) will be examined via a 2x2x2 design, in which 8 groups are created that all receive a different version of the intervention.

ELIGIBILITY:
Inclusion Criteria:

- 18 years old or older

Exclusion Criteria:

* Not Dutch-speaking
* Does not own a smartphone
* Does not have access to the internet
* Is not able to be physically active/non-sedentary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in objective physical activity (PA) | Baseline, 5 weeks, 3 months, 1 year
  Change in amount of total physical activity and moderate-to-vigorous physical activity, measured via accelerometers
Change in objective sedentary behaviour | Baseline, 5 weeks, 3 months, 1 year
  Change in amount of total sitting time, measured via accelerometers
Change in self-reported physical activity (PA) | Baseline, 5 weeks, 3 months, 1 year
  Change in amount of total physical activity and moderate-to-vigorous physical activity, measured via the International Physical Activity Questionnaire (IPAQ)
Change in self-reported sedentary behaviour | Baseline, 5 weeks, 3 months, 1 year
  Change in amount of total sitting time, measured via the last 7-days sedentary behaviour self-report questionnaire (SIT-Q-7d)

SECONDARY OUTCOMES:
Change in self-efficacy | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Change in amount of self-efficacy to change behaviour, measured via 3 validated items (questionnaire)
Change in motivation | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Change in amount of motivation to change behaviour, measured via 3 validated items (questionnaire)
Change in outcome expectancies | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Outcome expectancies regarding the behaviour change, measured via 3 validated items (questionnaire)
Change in risk perception | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Risk perception about the behaviour, measured via 3 validated items (questionnaire)
Change in intention | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Amount of intention to change behaviour, measured via 3 validated items (questionnaire)
Change in action planning | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Amount of action planning for behaviour change, measured via 3 validated items (questionnaire)
Change in coping planning | Baseline, 1 week, 3 weeks, 5 weeks, 3 months, 1 year
  Amount of coping planning for behaviour change, measured via 3 validated items (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Ilse De Bourdeaudhuij, Professor, Principal Investigator — University Ghent; Geert Crombez, Professor, Principal Investigator — University Ghent; Maïté Verloigne, PostDoc, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroe H, Carlier S, Van Dyck D, De Backere F, Crombez G. Towards more personalized digital health interventions: a clustering method of action and coping plans to promote physical activity. BMC Public Health. 2022 Dec 12;22(1):2325. doi: 10.1186/s12889-022-14455-4. PMID 36510181
- [Derived] Schroe H, Crombez G, De Bourdeaudhuij I, Van Dyck D. Investigating When, Which, and Why Users Stop Using a Digital Health Intervention to Promote an Active Lifestyle: Secondary Analysis With A Focus on Health Action Process Approach-Based Psychological Determinants. JMIR Mhealth Uhealth. 2022 Jan 31;10(1):e30583. doi: 10.2196/30583. PMID 35099400
- [Derived] Schroe H, Van Dyck D, De Paepe A, Poppe L, Loh WW, Verloigne M, Loeys T, De Bourdeaudhuij I, Crombez G. Which behaviour change techniques are effective to promote physical activity and reduce sedentary behaviour in adults: a factorial randomized trial of an e- and m-health intervention. Int J Behav Nutr Phys Act. 2020 Oct 7;17(1):127. doi: 10.1186/s12966-020-01001-x. PMID 33028335
- [Derived] Schroe H, Van der Mispel C, De Bourdeaudhuij I, Verloigne M, Poppe L, Crombez G. A factorial randomised controlled trial to identify efficacious self-regulation techniques in an e- and m-health intervention to target an active lifestyle: study protocol. Trials. 2019 Jun 10;20(1):340. doi: 10.1186/s13063-019-3456-7. PMID 31182147